CLINICAL TRIAL: NCT02896192
Title: An Open-Label, 1-Year Trial, Including a Double-Blind Placebo-Controlled Withdrawal Period, of Setmelanotide (RM-493), a Melanocortin 4 Receptor (MC4R) Agonist, in Early Onset POMC Deficiency Obesity Due to Bi-Allelic Loss-of-Function POMC or PCSK1 Genetic Mutation
Brief Title: Setmelanotide for the Treatment of Early-Onset Pro-Opiomelanocortin (POMC) Deficiency Obesity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RM-493-012; 2016-002320-83 (EudraCT Number)
Record Dates: First submitted 2016-08-18; First posted 2016-09-12 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Pro-opiomelanocortin (POMC) Deficiency Obesity
Keywords: POMC deficiency obesity; PCSK1 deficiency obesity; Setmelanotide; RM-493; Obesity; Melanocortin 4 receptor; MC4R pathway
MeSH Terms: conditions — Obesity | interventions — setmelanotide

STUDY DESIGN:
Intervention Model Description: Open-label with an 8 week Double-Blind Placebo-Controlled Withdrawal Period
Masking Description: During the 8 week double-blind placebo-controlled withdrawal period, participants received 4 weeks of daily setmelanotide and 4 weeks of daily placebo. Participants, investigators, and sites remained blinded as to when placebo treatment was administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Setmelanotide (Experimental): Participants received titrated doses of setmelanotide once daily, by subcutaneous (SC) injection during titration period for 2 - 12 weeks. Thereafter, participants continued setmelanotide at their specific therapeutic dose for an additional 10 weeks during the open label treatment period. Participants who achieved at least a 5 kilograms (kg) weight loss (or at least 5% weight loss if baseline body weight was <100 kg) at the end of the open label treatment period, continued into the 8-week double-blind withdrawal period and received 4 weeks setmelanotide and 4 weeks placebo. Following the withdrawal period, participants entered open label treatment period and received setmelanotide to complete approximately 52 weeks (~1 year) of treatment at a therapeutic dose.
  Interventions: Drug: Setmelanotide; Drug: Placebo

INTERVENTIONS:
Drug: Setmelanotide — Once daily SC injection
  Other Names: RM-493
Drug: Placebo — Once daily SC injection

SUMMARY:
To demonstrate statistically significant and clinically meaningful effects of setmelanotide on percent body weight change in participants with pro-opiomelanocortin (POMC) deficiency or proprotein convertase subtilisin/kexin type 1 (PCSK1) deficiency obesity due to rare biallelic or loss-of function mutations at the end of 1 year of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Bi-allelic, homozygous or compound heterozygous (a different gene mutation on each allele) genetic status for either the POMC or PCSK1 genes, with the loss-of-function (LOF) variant for each allele conferring a severe obesity phenotype.
2. Age 6 years and above.
3. If adult age ≥ 18 years, obesity with body mass index (BMI) ≥ 30 kilograms per square meter (kg/m^2); if child or adolescent, obesity with BMI ≥ 95th percentile for age on growth chart assessment.
4. Study participant and/or parent or guardian is able to communicate well with the investigator, to understand and comply with the requirements of the study, and be able to understand and sign the written informed consent/assent, after being informed about the study.
5. Female participants of child-bearing potential must agree to use contraception as outlined in the protocol. Female participants of non-childbearing potential, defined as surgically sterile (status post-hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months (and confirmed with a screening follicular stimulating hormone [FSH] level in the post-menopausal lab range), or have delayed pubertal development and failure to have achieved menarche, do not require contraception during the study.
6. Male participants with female partners of childbearing potential must agree to a double barrier method if they become sexually active during the study. Male participants must not donate sperm during and for 90 days following their participation in the study.

Exclusion Criteria:

1. Recent intensive (within 2 months) diet and/or exercise regimen with or without the use of weight loss agents, including herbal medications, that has resulted in weight loss or weight stabilization. Participants may be reconsidered approximately 1 month after cessation of such intensive regimens.
2. Prior gastric bypass surgery resulting in >10% weight loss durably maintained from the baseline pre-operative weight with no evidence of weight regain.
3. Diagnosis of schizophrenia, bipolar disorder, personality disorder or other Diagnostic and Statistical Manual of Mental Disorders (DSM-III) disorders that the investigator believes will interfere significantly with study compliance.
4. A Patient Health Questionnaire-9 (PHQ-9) score of ≥ 15.
5. Any suicidal ideation of type 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS). Any lifetime history of a suicide attempt, or any suicidal behavior in the last month.
6. Current, clinically significant pulmonary, cardiac, or oncologic disease.
7. History of significant liver disease or liver injury, or current liver assessment for a cause of abnormal liver tests (as indicated by abnormal liver function tests, alanine transaminase [ALT], aspartate transaminase [AST], alkaline phosphatase, or serum bilirubin [> 2.0 x upper limit of normal (ULN) for any of these tests]) for an etiology other than non-alcoholic fatty liver disease (NAFLD). Thus, any underlying etiology besides NAFLD, including diagnosed non-alcoholic steatohepatitis (NASH), other causes of hepatitis, or history of hepatic cirrhosis will be exclusionary, but the presence of NAFLD would not be exclusionary.
8. History or presence of impaired renal function as indicated by clinically significant abnormal creatinine, blood urea nitrogen (BUN), or urinary constituents (e.g., albuminuria) or moderate to severe renal dysfunction as defined by the Cockcroft Gault equation < 30 mL/min.
9. History or close family history (parents or siblings) of skin cancer or melanoma, or participant history of ocular-cutaneous albinism.
10. Significant dermatologic findings relating to melanoma or pre-melanoma skin lesions, determined as part of a screening comprehensive skin evaluation performed by a qualified dermatologist.
11. Participant is, in the opinion of the study investigator, not suitable to participate in the study.
12. Participation in any clinical study with an investigational drug/device within 3 months prior to the first day of dosing.
13. Significant hypersensitivity to study drug.
14. Inability to comply with every day (QD) injection regimen.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, MD, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (7):
- Honor Health Research Institute, Scottsdale, Arizona, United States
- UZ Gent, Ghent, Belgium
- Peel Memorial Hospital, Brampton, Ontario, Canada
- Institute of Cardiometabolism and Nutrition / Hopital de la Pitié-Salpêtrière, Paris, France
- Charité Campus Virchow-Klinikum / Institute for Experimental Pediatric Endocrinology, Berlin, Germany
- Hospital Universitario Niño Jesús, Madrid, Spain
- University of Cambridge Metabolic Research Laboratories, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clement K, van den Akker E, Argente J, Bahm A, Chung WK, Connors H, De Waele K, Farooqi IS, Gonneau-Lejeune J, Gordon G, Kohlsdorf K, Poitou C, Puder L, Swain J, Stewart M, Yuan G, Wabitsch M, Kuhnen P; Setmelanotide POMC and LEPR Phase 3 Trial Investigators. Efficacy and safety of setmelanotide, an MC4R agonist, in individuals with severe obesity due to LEPR or POMC deficiency: single-arm, open-label, multicentre, phase 3 trials. Lancet Diabetes Endocrinol. 2020 Dec;8(12):960-970. doi: 10.1016/S2213-8587(20)30364-8. Epub 2020 Oct 30. PMID 33137293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled into the pivotal cohort (10 participants) or supplemental cohort (5 participants).
  Pivotal cohort: Set of participants under study constituted a collection of detailed clinical case reports with a comprehensive baseline and past medical history assessment and complete clinical efficacy, safety and laboratory evaluations conducted for each participant.
  Supplemental cohort: Any additional participants enrolled were included in supplemental cohort.
Pre-assignment Details: At screening, a blood sample was obtained for genotyping for mechanisms considered to be possibly related to the safety or efficacy response to the study medication (e.g., other obesity related genes). Complete physical, relevant bloodwork, and other standard assessments were performed.
Period: Titration Period (2 to 12 Weeks)
Arm/Group | Setmelanotide
Started | 15
Treated | 15
Completed | 15
Not Completed | 0
Period: Open-Label Period (10 Weeks)
Arm/Group | Setmelanotide
Started | 15
Completed | 13
Not Completed | 2
Not completed — Lack of Efficacy | 1
Not completed — Protocol Violation | 1
Period: Double-Blind Withdrawal Period (8 Weeks)
Arm/Group | Setmelanotide
Started | 13
Completed | 13
Not Completed | 0
Period: Open-Label Period (32 Weeks)
Arm/Group | Setmelanotide
Started | 13
Completed | 12
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAS) Population consisted of participants who received any of the study drug injections and had at least one post-dose safety assessment.
Groups:
- Setmelanotide: Participants received titrated doses of setmelanotide once daily, by SC injection during titration period for 2 - 12 weeks. Thereafter, participants continued setmelanotide at their specific therapeutic dose for an additional 10 weeks during the open label treatment period. Participants who achieved at least a 5 kg weight loss (or at least 5% weight loss if baseline body weight was <100 kg) at the end of the open label treatment period, continued into the 8-week double-blind withdrawal period and received 4 weeks setmelanotide and 4 weeks placebo. Following the withdrawal period, participants entered open label treatment period and received setmelanotide to complete approximately 52 weeks (~1 year) of treatment at a therapeutic dose.
Arm/Group | Setmelanotide
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.20 (7.02)
Age, Customized [Count of Participants; unit: Participants]
  < 12 years | 5
  ≥ 12 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 1
  Belgium | 2
  United States | 1
  France | 2
  Germany | 7
  Spain | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Reached ≥10% Weight Loss Threshold After 1 Year (Pivotal Cohort)
Description: The percentage of participants who met the ≥ 10% weight loss threshold after approximately Week 52 (~1 year) of treatment were analyzed.
Time Frame: Week 52
Population: Full Analysis Set (FAS) population included participants who received any of the study drug injections and had at least one baseline assessment (included those who did and did not demonstrate ≥ 5 kg weight loss or 5% of body weight if weight was < 100 kg at baseline over the 12-week open-label treatment period, and proceeded into the double-blind, placebo-controlled withdrawal period). Participants in pivotal cohort were included in the analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Setmelanotide (Entire Study): Participants received setmelanotide once daily by SC injection for approximately 52 weeks (~ 1 year).
Arm/Group | Setmelanotide (Entire Study)
Number analyzed (Participants) | 10
percentage of participants | 80.0 [49.31 to 96.32]
Statistical Analysis 1: Comparison: Setmelanotide (Entire Study); Test type: Other; p < 0.0001, Exact binomial test — One-sided p-value obtained from exact binomial test, testing that at least 5% of participants in the population of interest would achieve 10% weight loss; CI

2. Secondary Outcome: Percentage of Participants Who Reached ≥10% Weight Loss Threshold After 1 Year (Pivotal + Supplemental Cohort)
Description: as for outcome 1
Time Frame: Week 52
Population: FAS Population. Participants in pivotal and supplemental cohort were included in the analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Setmelanotide (Entire Study)
Number analyzed (Participants) | 14
percentage of participants | 85.7 [61.46 to 97.40]
Statistical Analysis 1: Comparison: Setmelanotide (Entire Study); Test type: Other; p < 0.0001, Exact binomial test — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Mean Percent Change From Baseline in Body Weight at Week 52
Description: The mean percent change from baseline in body weight at 52 weeks was analyzed.
Time Frame: Baseline, Week 52
Population: Designated Use Set (DUS) analysis population consisted of participants who received any of the study drug injections, demonstrated ≥ 5 kg weight loss or 5% of body weight if weight was <100 kg at baseline over the 12-week open-label treatment period, and proceeded into the double-blind, placebo-controlled withdrawal period. Participants in pivotal and supplemental cohort were included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Setmelanotide (Entire Study)
Number analyzed (Participants) | 13
percent change | -25.83 (9.721)
Statistical Analysis 1: Comparison: Setmelanotide (Entire Study); Model based summary statistics from longitudinal mixed analysis of variance model with fixed effect for visit, baseline body weight and random effect for participant, one sided p-value from model; Test type: Other; p < 0.0001, Longitudinal mixed analysis of variance; Least Squares Mean = -25.73, 90% CI 2-sided [-28.49 to -22.98]

4. Secondary Outcome: Mean Percent Change From Baseline in Hunger Score (Worst "Most" Hunger in 24 Hours) at Week 52
Description: The mean percent change in hunger scores for participants ≥12 years of age with leptin receptor (LEPR) deficiency obesity in treatment with setmelanotide was evaluated. Hunger score ranged from 0 - 10 on a Likert-type scale; 0 = not hungry at all and 10 = hungriest possible. On the Daily Hunger Questionnaire, each of the 3 items (average hunger, most/worst hunger, and morning hunger) was scored separately and averaged on a weekly basis. The weekly average hunger score of the daily worst (most) hunger score in 24 hours is the hunger score used to assess this study endpoint.
Time Frame: Baseline, Week 52
Population: Participants in the DUS population with available data were analyzed. Participants in pivotal and supplemental cohort were included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Setmelanotide (Entire Study)
Number analyzed (Participants) | 7
percent change | -27.1 (28.11)
Statistical Analysis 1: Comparison: Setmelanotide (Entire Study); Model based summary statistics from longitudinal mixed analysis of variance model with fixed effect for week, baseline daily hunger score and random effect for participant, one sided p-value from model; Test type: Other; p = 0.0005, Longitudinal mixed analysis of variance; Least Squares Mean = -27.77, 90% CI 2-sided [-40.58 to -14.96]

5. Secondary Outcome: Percentage of Participants Who Achieved at Least 25% Improvement in Daily Hunger From Baseline
Description: The percentage of participants (≥12 years of age) achieving a ≥25% improvement from baseline in hunger score at Week 52 (i.e., after treatment with setmelanotide for 52 weeks at the therapeutic dose) was assessed. Hunger ranged from 0 - 10 on a Likert-type scale; 0 = not hungry at all and 10 = hungriest possible. On the Daily Hunger Questionnaire, each of the 3 items (average hunger, most/worst hunger, and morning hunger) was scored separately and averaged on a weekly basis. The weekly average hunger score of the daily worst (most) hunger score in 24 hours is the hunger score used to assess this study endpoint.
Time Frame: Baseline, Week 52
Population: Participants in the FAS population with available data were analyzed. Participants in pivotal and supplemental cohort were included in the analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Setmelanotide (Entire Study)
Number analyzed (Participants) | 8
percentage of participants | 50.0 [19.29 to 80.71]
Statistical Analysis 1: Comparison: Setmelanotide (Entire Study); Test type: Other; p = 0.0004, Exact binomial test — One-sided p-value obtained from exact binomial test, testing that ≥ 5% of participants in the population of interest would achieve ≥ 25% improvement in daily hunger score

6. Secondary Outcome: Absolute Change From Baseline in Waist Circumference at Week 52
Description: Waist circumference (centimeters) was measured according to the National Heart, Lung, and Blood Institute (NHLBI) criteria. Waist circumference was measured when participants were fasting at approximately the same time at each visit. The absolute change from baseline in waist circumference was assessed.
Time Frame: Baseline, Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Setmelanotide (Entire Study)
Number analyzed (Participants) | 13
centimeters
  Baseline | 115.48 (17.920)
  Change at Week 52: number analyzed (Participants) | 11
  Change at Week 52 | -17.51 (9.112)
Statistical Analysis 1: Comparison: Setmelanotide (Entire Study); Model based summary statistics from longitudinal mixed analysis of variance model with fixed effect for visit, baseline waist circumference and random effect for participant, one sided p-value from model; Test type: Other; p < 0.0001, Longitudinal mixed analysis of variance; Least Squares Mean = -18.1, 90% CI 2-sided [-21.27 to -14.88]

7. Secondary Outcome: Absolute Change in Body Weight (Reversal of Weight Loss) During Double-Blind Placebo-Controlled Withdrawal Period
Description: A comparison of weight change was evaluated during the 8 week placebo-controlled withdrawal period for each participant, during which each participant received 4 weeks of placebo and 4 weeks active therapy in a blinded fashion.
Time Frame: Baseline, 8-week withdrawal period (up to ~Week 20)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kilograms
Groups:
- Setmelanotide (Double-Blind): Participants received setmelanotide once daily by SC injection for 4 weeks and placebo matched to setmelanotide for 4 weeks during the double-blind placebo controlled withdrawal period.
Arm/Group | Setmelanotide (Double-Blind)
Number analyzed (Participants) | 11
kilograms
  Change after 4 weeks of therapy: Setmelanotide | -2.8 (2.41)
  Change after 4 weeks of therapy: Placebo | 6.2 (3.87)

8. Secondary Outcome: Absolute Score in Daily Hunger Reduction During the Double-Blind Placebo-Controlled Withdrawal Period
Description: The absolute score in daily hunger during the double-blind placebo-controlled withdrawal period (≥12 Years of Age) was assessed. Hunger ranged from 0 - 10 on a Likert-type scale; 0 = not hungry at all and 10 = hungriest possible. On the Daily Hunger Questionnaire, each of the 3 items (average hunger, most/worst hunger, and morning hunger) was scored separately and averaged on a weekly basis. The weekly average hunger score of the daily worst (most) hunger score in 24 hours is the hunger score used to assess this study endpoint. Lower scores represent lower hunger, higher scores represent greater hunger.
Time Frame: 8-week withdrawal period (up to ~Week 20)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Setmelanotide (Double-Blind)
Number analyzed (Participants) | 7
units on a scale
  Setmelanotide | 4.5 (2.57)
  Placebo | 6.7 (2.22)

9. Secondary Outcome: Mean Percent Change From Baseline in Body Mass Index (BMI) at Week 52
Description: The mean percent change from baseline in BMI was assessed.
Time Frame: Baseline, Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Setmelanotide (Entire Study)
Number analyzed (Participants) | 11
percent change | -27.32 (8.971)
Statistical Analysis 1: Comparison: Setmelanotide (Entire Study); Model based summary statistics from longitudinal mixed analysis of variance model with fixed effect for week, baseline BMI and random effect for participant, one sided p-value from model; Test type: Other; p < 0.0001, Longitudinal mixed analysis of variance; Least Squares Mean = -27.4, 90% CI 2-sided [-30.60 to -24.29]

10. Secondary Outcome: Area Under the Curve (AUC) Change From Baseline in Oral Glucose, Assessed by the Oral Glucose Tolerance Test (OGTT)
Description: The AUC change from baseline for the OGTT was assessed. The AUC was calculated by the linear trapezoidal method and includes pre-dose and post-dose assessments. At each visit, oral glucose was captured pre-meal, and post-meal at the following times: 30 minutes, 60 minutes, 90 minutes, and 120 minutes. OGTT was not performed for participants with a diagnosis of Type 1 or Type 2 diabetes.
Time Frame: Baseline, Week 52
Population: Participants in the SAS population with available data were analyzed. Participants in pivotal and supplemental cohort were included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes*millimoles/liter (min*mmol/L)
Arm/Group | Setmelanotide (Entire Study)
Number analyzed (Participants) | 13
minutes*millimoles/liter (min*mmol/L)
  Baseline | 951.900 (464.9342)
  Change at Week 52: number analyzed (Participants) | 8
  Change at Week 52 | -35.284 (442.6334)

11. Secondary Outcome: Change From Baseline in Serum Glucose at Week 52
Description: Change from baseline in serum glucose at Week 52 was assessed.
Time Frame: Baseline, Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Setmelanotide (Entire Study)
Number analyzed (Participants) | 15
mmol/L
  Baseline | 6.606 (5.0024)
  Change at Week 52: number analyzed (Participants) | 10
  Change at Week 52 | -1.527 (1.9374)

ADVERSE EVENTS:
Time Frame: From first dose up to ~30 days after last dose of study drug (Up to ~ 1 year)
Description: SAS population. Participants in pivotal and supplemental cohort were included. Adverse events were analyzed for participants in the setmelanotide group (including the placebo withdrawal period) and adverse event data were not collected separately by period (or during placebo withdrawal) since all participants were exposed to setmelanotide.
Arm/Group | Setmelanotide
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 6/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Setmelanotide (N=15)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Major Depression (Psychiatric disorders) | 1 (1)
Panic Attack (Psychiatric disorders) | 1 (1)
Adrenocortical Insufficiency Acute (Endocrine disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Setmelanotide (N=15)
Haematoma (Vascular disorders) | 1 (1)
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7)
Multiple Allergies (Immune system disorders) | 1 (1)
Injection Site Erythema (General disorders) | 12 (59)
Injection Site Oedema (General disorders) | 9 (29)
Injection Site Pruritus (General disorders) | 9 (20)
Fatigue (General disorders) | 6 (7)
Chills (General disorders) | 3 (4)
Injection Site Pain (General disorders) | 4 (4)
Asthenia (General disorders) | 3 (3)
Injection Site Bruising (General disorders) | 3 (3)
Pyrexia (General disorders) | 2 (3)
Injection Site Induration (General disorders) | 2 (2)
Hyperthermia (General disorders) | 1 (1)
Injection Site Discolouration (General disorders) | 1 (1)
Injection Site Nodule (General disorders) | 1 (1)
Temperature Intolerance (General disorders) | 1 (1)
Thirst (General disorders) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 2 (3)
Depressed Mood (Psychiatric disorders) | 2 (2)
Restlessness (Psychiatric disorders) | 2 (2)
Sleep Disorder (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1)
Spontaneous Penile Erection (Reproductive system and breast disorders) | 2 (5)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Erection Increased (Reproductive system and breast disorders) | 1 (1)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 1 (1)
Blood Bilirubin Increased (Investigations) | 1 (1)
Blood Potassium Decreased (Investigations) | 1 (1)
Blood Thyroid Stimulating Hormone Increased (Investigations) | 1 (1)
Blood Uric Acid Increased (Investigations) | 1 (1)
International Normalised Ratio Increased (Investigations) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 1 (1)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 8 (14)
Disturbance in Attention (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Parosmia (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (5)
Nausea (Gastrointestinal disorders) | 8 (18)
Vomiting (Gastrointestinal disorders) | 8 (17)
Abdominal Pain (Gastrointestinal disorders) | 4 (10)
Diarrhoea (Gastrointestinal disorders) | 5 (7)
Dry Mouth (Gastrointestinal disorders) | 4 (5)
Lip Dry (Gastrointestinal disorders) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 15 (24)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (4)
Dry Skin (Skin and subcutaneous tissue disorders) | 4 (4)
Rash Papular (Skin and subcutaneous tissue disorders) | 2 (2)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1)
Perioral Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle Contracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Cortisol Deficiency (Endocrine disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Hypovitaminosis (Metabolism and nutrition disorders) | 1 (1)
Selenium Deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin A Deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 7 (16)
Gastroenteritis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pharyngitis Streptococcal (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Viral Infection (Infections and infestations) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
There was no planned comparison to a randomized placebo group given the rarity of monogenic POMC deficiency obesity. To provide support in assessing setmelanotide treatment in this open-label single-arm trial design, individual participants were evaluated during a double-blind placebo-controlled withdrawal phase in which participants served as their own control to assess effects on weight and reported hunger scores.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information regarding setmelanotide supplied by Rhythm to the investigator is privileged and confidential information. The investigator agrees to use this information to accomplish the study and will not use it for other purposes without consent from Rhythm. The information obtained from the clinical study will be used towards the development of setmelanotide and may be disclosed to regulatory authority(ies), other investigators, corporate partners, or consultants as required.

DOCUMENTS (2):
  • Study Protocol (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT02896192/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/92/NCT02896192/SAP_001.pdf